CLINICAL TRIAL: NCT04419532
Title: A Phase 1, First In Human Study of DS-1055a in Subjects With Relapsed or Refractory Locally Advanced or Metastatic Solid Tumors
Brief Title: A Study Evaluating DS-1055a in Participants With Relapsed or Refractory Locally Advanced or Metastatic Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DS1055-A-J101
Record Dates: First submitted 2020-06-03; First posted 2020-06-05 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Solid Tumor; Advanced Cancer; Metastatic Solid Tumor
Keywords: Solid Tumor; Advanced Cancer; Metastatic Solid Tumor; DS-1055a
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dose Escalation (DS-1055a) (Experimental): Participants will be enrolled into groups with each group receiving an increased dose from the previous group as safety assessments permit in order to determine the optimal dose for safety and tolerability.
  Interventions: Drug: DS-1055a

INTERVENTIONS:
Drug: DS-1055a — Administered as an intravenous infusion on Day 1 of every 21-day cycle following low dose administration(s) in priming dose period.
  Infusion duration: 180 minutes for the first infusion, and if no infusion-related reaction, 120 minutes for subsequent infusions

SUMMARY:
The purpose of this study is to assess the safety and tolerability of DS-1055a in participants with relapsed or refractory locally advanced or metastatic solid tumors for which no standard treatment is available.

DETAILED DESCRIPTION:
This Phase 1, open-label, non-randomized, dose escalation, first-in-human study will assess the safety and tolerability of DS-1055a, determine the maximum tolerated dose of DS-1055a, pharmacokinetic (PK) properties of DS-1055a, and the incidence of anti-drug antibodies (ADAs) against DS-1055a and other antibodies.

ELIGIBILITY:
Inclusion Criteria:

* Has a histopathologically documented locally advanced or metastatic head and neck, gastric, esophageal cancer, non-small cell lung cancer, or melanoma. Participants with other types of solid tumors may be eligible following discussion with the Sponsor.
* Has a relapsed or refractory disease that is not amenable to curative standard therapy.
* Is 18 years of age or older.
* Has an Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0-1, with no deterioration for two weeks.
* Has a measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
* Has adequate organ function within 7 days before enrollment.
* Is able to provide written informed consent and is willing and able to comply with the protocol.

Exclusion Criteria:

* Has a concurrently active second malignancy, other than adequately treated non-melanoma skin cancers, in situ melanoma or in situ cervical cancer. Participants with history of the second malignancy have been disease-free for <3 years.
* Has a history of (non-infectious) interstitial lung disease (ILD) that required steroids, currently has ILD, or when suspected ILD cannot be ruled out by imaging at screening.
* Has a history of severe pulmonary compromise or requirement of supplemental oxygen within 6 months before enrollment.
* Has active hepatitis B or hepatitis C virus infection.
* Has received prior immunotherapy with a Grade 3 or higher, or any unresolved ≥Grade 2 immune-related adverse event.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-10-09 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with dose-limiting toxicities | 21 days of Cycle 1
  A dose-limiting toxicity (DLT) is defined as any treatment-emergent adverse event (TEAE) that occurs during the DLT evaluation period (21 days), excluding toxicities clearly related to disease progression or intercurrent illness or to concomitant medications or to concomitant procedures and is Grade 3 or above according to National Cancer Institute-Common Terminology Criteria for Adverse Events Version 5.0, with certain specified exceptions.
Number of participants with adverse events | Baseline up to approximately 3 years
  Adverse events were assessed using National Cancer Institute-Common Terminology Criteria for Adverse Events Version 5.0.

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | Priming Dose Cycle 1 Day 1 to Cycle 4 Day 1, and every 2 cycles from Cycle 4 to end of treatment, within approximately 2 years (each cycle is 21 days)
Time to Reach Maximum Plasma Concentration (Tmax) | Priming Dose Cycle 1 Day 1 to Cycle 4 Day 1, and every 2 cycles from Cycle 4 to end of treatment, within approximately 2 years (each cycle is 21 days)
Area Under the Plasma Concentration-Time Curve Up to Last Quantifiable Time (AUClast) and During Dosing Interval (AUCtau) | Priming Dose Cycle 1 Day 1 to Cycle 4 Day 1, and every 2 cycles from Cycle 4 to end of treatment, within approximately 2 years (each cycle is 21 days)
Minimum Observed Concentration (Ctrough) | Priming Dose Cycle 1 Day 1 to Cycle 4 Day 1, and every 2 cycles from Cycle 4 to end of treatment, within approximately 2 years (each cycle is 21 days)
The Incidence of Anti-Drug Antibodies (ADA) and Other Antibodies | From pre-treatment to follow-up visit (within approximately 2 years)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Leader, Study Director — Daiichi Sankyo
Locations (6):
- United States (2):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Cincinnati Cancer Center, Cincinnati, Ohio
- Princess Margaret Cancer Center, Toronto, Ontario, Canada
- Japan (3):
  - National Cancer Center Hospital, Chūōku
  - National Cancer Center Hospital East, Kashiwa
  - Cancer Institute Hospital of JFCR, Kōtoku

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) on completed studies and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Completed studies that has reached a global end or completion with all data set collected and analyzed, and for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents on completed clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/